CLINICAL TRIAL: NCT02058407
Title: A Randomised, Double-blind (Sponsor Unblind), Placebo-controlled, Two Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single or Repeat Doses of GSK2793660 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) and Food Effect of Single or Repeat Doses of GSK2793660 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug related AEs observed upon repeat dosing that with longer treatment duration could become worse. Required action on some biomarkers not observed.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 200186
Record Dates: First submitted 2014-01-09; First posted 2014-02-10 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Bronchiectasis
Keywords: food effect; pharmacokinetics; GSK2793660; FTIH; pharmacodynamics; safety
MeSH Terms: conditions — Bronchiectasis | interventions — GSK-2793660

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1- Part A (Experimental): This cohort will follow an interlocking design with Cohort 2 - Part A. Out of the 9 healthy subjects in this cohort, 3 subjects will receive placebo and 6 subjects will receive GSK2793660 according to randomization schedule in three single-dose study periods. Drug administration will be staggered over 2 days in each period. On Day 1, only 1 subject will receive GSK2793660 and 1 subject will receive placebo. The remaining subjects will be dosed on Day 2 of each treatment period assuming adequate safety from Day 1. Placebo administration and an escalation of GSK2793660 from 0.5 mg, to 3 mg, and 20 mg in the subsequent periods, will be done with a minimum washout period of 13 days between doses. If the target clinical dose is determined as being one of the doses administered to this cohort, they will have an additional study period for the administration of target clinical dose GSK2793660 following the standard Food and drug administration (FDA) high fat/high calorie meal.
  Interventions: Drug: GSK2793660 solution; Drug: GSK2793660 capsule; Drug: Placebo solution; Drug: Placebo capsule
- Cohort 2- Part A (Experimental): This cohort will follow an interlocking design with Cohort 1 - Part A. Out of the 9 healthy subjects in this cohort, 3 subjects will receive placebo and 6 subjects will receive GSK2793660 according to randomization schedule in three single-dose study periods. Drug administration will be staggered over 2 days in each period. On Day 1, only 1 subject will receive GSK2793660 and 1 subject will receive placebo. The remaining subjects will be dosed on Day 2 of each treatment period assuming adequate safety from Day 1. Placebo administration and an escalation of GSK2793660 from 1 mg, to 10 mg, and 50 mg in the subsequent periods, will be done with a minimum washout period of 13 days between doses. If the target clinical dose is determined as being one of the doses administered to this cohort, they will have an additional study period for the administration of target clinical dose GSK2793660 following the standard FDA high fat/high calorie meal.
  Interventions: Drug: GSK2793660 solution; Drug: GSK2793660 capsule; Drug: Placebo solution; Drug: Placebo capsule
- Cohort 3- Part B (Experimental): It is planned that up to two doses evaluated in Part A will be taken through to Part B. In this cohort, the lower dose (which will be the likely clinically efficacious dose) will be given for 14 days. The dosing frequency (once a day or twice daily) will be based on a review of the safety, tolerability, PK and PD data from Part A. It is planned that 10 subjects will receive GSK2793660 and 5 subjects will receive placebo. Subjects will be dosed on Day 1 and then on Days 3-15 (assuming once-daily dosing). If dosing is twice-daily, doses will be administered in the morning and evening from Day 1-14.
  Interventions: Drug: GSK2793660 capsule; Drug: Placebo capsule
- Cohort 4- Part B (Experimental): It is planned that up to two doses evaluated in Part A will be taken through to Part B. In this cohort, the higher dose (maximum tolerated or safe dose) will be given for 14 days. The dosing frequency (once a day or twice daily) will be based on a review of the safety, tolerability, PK and PD data from Part A. It is planned that 10 subjects will receive GSK2793660 and 5 subjects will receive placebo. Subjects will be dosed on Day 1 and then on Days 3-15 (assuming once-daily dosing). If dosing is twice-daily, doses will be administered in the morning and evening from Day 1-14. Cohort 4 will commence only after Cohort 3 is completed and data is reviewed. Also there will be no Cohort 4, if only one dose is to be evaluated in Part B.
  Interventions: Drug: GSK2793660 capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: GSK2793660 solution — Clear, colourless solution at a unit dose strength of 0.1 mg/mL, in a glass bottle
  Arms: Cohort 1- Part A; Cohort 2- Part A
Drug: GSK2793660 capsule — Size zero swedish orange capsule at a unit dose of 3 mg, 10 mg, 20 mg and 50 mg
Drug: Placebo solution — Matching placebo to GSK2793660 solution
  Arms: Cohort 1- Part A; Cohort 2- Part A
Drug: Placebo capsule — Matching placebo to GSK2793660 capsule

SUMMARY:
This study is the first administration of GSK2793660 to humans and will evaluate the safety, tolerability, PK and PD of single oral ascending doses of GSK2793660, and of repeat oral doses of GSK2793660 in healthy subjects. The study will comprise two parts (Part A and Part B). Part A will consist of two cohorts of subjects, each taking part in a three-way cross over study, with ascending doses of GSK2793660 and placebo. Available safety, PK and PD data will be reviewed before each dose escalation. This will be followed by a food-effect arm in the cohort that received what is deemed to be the target clinical dose. Part B is planned to consist of up to two cohorts of subjects, each taking part in one 14 day repeat dose study period. Subjects will be dosed on Day 1 and then on Days 3-15. It is planned that two doses will be evaluated. The dose(s) to be tested will be selected based on safety, PK, and PD from Part A. The study is intended to provide sufficient confidence in the safety profile of the molecule and information on target engagement to allow progression to further studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, and laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range, and which is not a part of an eligibility criterion, for the population being studied may be included only if the Investigator and GSK medical monitor consider the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures and outcome.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, removal of both ovaries or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >21.7 International units per liter (IU/L) and oestradiol <110 picomole per liter (pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods listed in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects with female partners of child-bearing potential must agree to use one of the approved contraception methods as detailed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight >=50 Kilogram (kg) and Body Mass Index (BMI) within the range 19.9-30.0 kg/meter square (m^2) (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Based on averaged QT duration corrected for heart rate by Fridericia's formula (QTcF) values of triplicate ECGs obtained over a brief recording period: Average QTcF <450 milliseconds (msec)
* Systolic blood pressure <=130 millimeters of mercury (mmHg) and diastolic blood pressure 80 mmHg based on average values of triplicate blood pressure readings obtained over a brief period.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* ECG finding of second or third degree heart block.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Urinary cotinine or exhaled breath carbon monoxide (CO) levels indicative of current smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period. Blood donation will not exceed 500 mL for the entire study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2793660 as assessed by vital signs in Part A and Part B | Part A: Screening (SCR), Day 1 (Pre-dose, 0.25 hours (h), 0.5 h, 1.5 h, 2 h, 3 h, 4 h, 12 h), Day 2 (24 h), Day 3 (48 h), Day 4 (72 h) in each period and at follow-up (7-14 days post last dose); Part B: SCR, Day 1 to Day 18 and at follow-up
  Vital sign measurements will include systolic and diastolic blood pressure, pulse rate, respiratory rate and oral body temperature
Safety and tolerability of GSK2793660 as assessed by cardiac telemetry in Part A and Part B | Part A: From 1 h pre-dose on Day 1 until 24 h post dose on Day 2 in each period. Part B: From 1 h prior to dosing on Day 3 until pre-dose on Day 5
  Continuous cardiac telemetry will be performed in Part A and Part B of the study
Safety and tolerability of GSK2793660 as assessed by electrocardiograms (ECGs) in Part A and Part B | Part A: SCR, Day 1 (Pre-dose, 0.25 h, 0.5 h, 1.5 h, 2 h, 3 h, 4 h, 12 h), Day 2 (24 h), Day 3 (48 h), Day 4 (72 h) in each period and at follow-up (7-14 days post last dose); Part B: SCR, Day 1 to Day 18 and at follow-up
  Cardiac safety will be assessed by 12-lead ECGs
Safety and tolerability of GSK2793660 as assessed by laboratory data in Part A and Part B | Part A: SCR, Day -1, Day 1 (8 h), Day 2 (24 h), Day 4 (72 h) in each period and at follow-up (7-14 days post last dose); Part B: SCR, Day -1, Day 2, Day 4, Day 10, Day 15, Day 18 and at follow-up
  Laboratory assessments will include hematology, clinical chemistry and urinalysis parameters
Safety and tolerability of GSK2793660 as assessed by adverse events (AEs) in Part A and Part B | Part A: Approximately 22- 24 weeks. Part B: Approximately 9 weeks

SECONDARY OUTCOMES:
Composite of PK parameters for GSK2793660 in Part A and Part B | Part A: Pre-dose, 0.25, 0.5, 1.5, 2, 3, 6, 8, 12, 16, 24, 30, 48 and 72 h; Part B: Days 1 and 15 (Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 6, 8 and 12 h), Days 2 and 16 (16, 24 and 30 h), Days 3 and 17 (48 h), Day 18 (72 h), Days 4, 7, 9, 11, 13 (pre-dose)
  PK parameters for GSK2793660 in plasma will include: area under the plasma concentration-time curve (AUC[0-t], AUC[0-infinity]), maximum observed plasma concentration (Cmax), time to Cmax (Tmax), apparent terminal phase half-life (T1/2).
To evaluate biomarker activity following oral administration of GSK2793660 in Part A and Part B | Part A: Pre-dose, 1 h, 2 h, 3 h, 6 h, 8 h, 12 h, 24 h, 30 h, 48 h, 72 h, 144 h in each period; Part B: Day 1 and Day 15 (Pre-dose, 1 h, 3 h, 6 h, 8 h and 12 h), Day 2 and Day 16 (24 h and 30 h), Day 3 and Day 17 (48 h), Day 18 (72 h)
  Blood biomarkers that will provide information on target engagement and downstream PD activity will be assessed. Biomarker endpoints including, but not limited to, cathepsin C enzyme activity in whole blood following single dose administration. Neutrophil serine protease activity (i.e. neutrophil elastase, cathepsin G, proteinase 3 [PR3]) following repeat dose administration. Other endpoints may include LL37 in cell extracts and surface expression of PR3 on neutrophils following repeat dose administration.
Effect of food on PK of GSK2793660 in Part A | Pre-dose, 0.25, 0.5, 1.5, 2, 3, 6, 8, 12, 16, 24, 30, 48 and 72 h
  PK parameters for GSK2793660 in plasma will include: AUC(0-t), AUC(0-infinity), Cmax, Tmax, and T1/2.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Miller BE, Mayer RJ, Goyal N, Bal J, Dallow N, Boyce M, Carpenter D, Churchill A, Heslop T, Lazaar AL. Epithelial desquamation observed in a phase I study of an oral cathepsin C inhibitor (GSK2793660). Br J Clin Pharmacol. 2017 Dec;83(12):2813-2820. doi: 10.1111/bcp.13398. Epub 2017 Sep 20. PMID 28800383
- See also: Results for study 200186 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200186?search=study&search_terms=200186#rs